CLINICAL TRIAL: NCT05670301
Title: Flemish Joint Effort for Biomarker PRofiling in Inflammatory Systemic Diseases
Acronym: FEBRIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Hospital, Antwerp (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Universitair Ziekenhuis Brussel (Other); Jessa Hospital (Other); Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-11141
Record Dates: First submitted 2022-01-31; First posted 2023-01-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Autoinflammatory Disease; Autoimmune Diseases; Inflammation
MeSH Terms: conditions — Autoimmune Diseases; Inflammation

STUDY DESIGN:
Masking Description: Pseudonymisation of samples and clinical data for the investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Cytokine assessment
  Interventions: Diagnostic Test: cytokine and lipidomic profiling

INTERVENTIONS:
Diagnostic Test: cytokine and lipidomic profiling — * FEBRIS Cytokine Profile Assay (quantification of inflammatory cytokines)
  * Serum amyloid A
  * Biobanking of leftover sample for future analyses and specific immunofunctional assay in selected cases
  * Lipidomics

SUMMARY:
A multi-centre, prospective study to study cytokine profiles and other potential disease-specific biomarkers in patients with presumed or confirmed diseases of systemic inflammation

The goal of this prospective, observational study is to describe the longitudinal evolution of blood cytokine profiles in patients with presumed or confirmed diseases of systemic inflammation

The main questions it aims to answer are:

* What are the differences and similarities in blood cytokines between different patients and groups presenting symptoms of systemic inflammatory conditions?
* How is the cytokine profile of individual patients evolving over time and what is the effect of different therapeutics?
* Is cytokine profiling a valuable tool to diagnose and follow-up on patients with systemic inflammatory conditions?

Participants will be asked to give an additional blood volume for research purposes when blood sampling is performed for routine clinical purposes. A subset of patients (those initiated on biologicals) will also be asked to complete questionnaires.

Researchers will compare the blood cytokines profiles between the different groups of systemic inflammatory conditions and with healthy individuals.

DETAILED DESCRIPTION:
FEBRIS is a prospective, observational and multi-centric study involving 5 hospitals in Flanders, Belgium.

In this study, the researchers will us ehe FEBRIS Cytokine Profile Assay, which is a multiplex assay measuring pro- and anti-inflammatory cytokines in the blood of subjects. It has been developed in a retrospective cohort of human patients presenting systemic inflammatory disorders.

With this study, the researchers aim to prospectively validate the use of this assay in a cohort of patients that present signs reminiscent of systemic inflammation, including patients with antoinflammatory conditions, autoimmune disorders, hyperinflammatory syndromes (e.g. hemophagocytic lymphohistiocytosis and macrophage activation syndrome) and systemic infection. In parallel, serum amyloid A will be quantified in all patients. Lipidomics will be performed on patients with sufficient leftover sample. The researchers will integrate the data from these assays with clinical parameters at baseline and during follow-up to correlate markers with the clinical or genetic diagnosis, prognosis and effect of different therapeutics.

Patients fulfilling the inclusion criteria are eligible for longitudinal blood sampling (every 3-6 months) during the study period (maximum of 4 years). Additional clotted blood will only be collected when a blood sample for routine clinical purposes is performed.

In addition, patients initiated on biological therapeutics will be asked to complete questionnaires regarding health-related quality of life to document outcome and improve rational and cost-efficient use of additional investigations and treatment.

ELIGIBILITY:
Inclusion Criteria:

An individual who meets any of the following criteria can be eligible for participation in this study:

1. Child or adult
2. Written informed consent
3. Suspected or confirmed disease with systemic inflammation (acute, chronic and/or recurrent), these include:

   1. Autoinflammatory diseases (AID), including among others: systemic onset juvenile idiopathic arthritis (sJIA), familial mediterranean fever (FMF), mevalonate kinase deficiency (Hyper IgD syndrome), TNF receptor-associated periodic syndrome (TRAPS), familial Cold Autoinflammatory Syndrome (CAPS), type 1 interferonopathies,…
   2. Autoimmune diseases (AI), including among others: systemic lupus erythematosus (SLE), juvenile dermatomyositis (JDM), rheumatoid arthritis (RA),…
   3. Hyperinflammatory diseases, including among others: hemophagocytic lymphohistiocytosis (HLH), macrophage activation syndrome (MAS), infection-related cytokine storm (e.g. in the setting of COVID-19)
   4. Other unidentified or not yet identified systemic inflammatory conditions
4. Blood sample for diagnostic purposes is planned and possibility to acquire additional blood volume

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Confirmed localized infection and/or good response to first-line antibiotic treatment
2. Confirmed malignancy

Besides the above mentioned patients, volunteers that meet the requirements as a healthy individual are eligible for inclusion as controls.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of inflammatory cytokines (interleukin (IL) 1 beta, IL-1RA, IL-6, IL-18, tumor necrosis factor (TNF) alpha, CXCL9 and CXCL10) on serum of patients | full study period (up to 48 months)
  On the sera of patients, the FEBRIS Cytokine Profile Assay will be performed.
  The FEBRIS Cytokine Profile Assay is a multiplex panel of inflammatory cytokines (interleukin (IL) 1 beta, IL-1RA, IL-6, IL-18, tumor necrosis factor (TNF) alpha, CXCL9 and CXCL10) that will be assessed by Meso Scale Discovery (MSD) technology. The concentration of cytokines will be quantified in pg/ml.
  Sera will be analyzed upon entry in the study and during follow-up (minimum interval of 3 months between samples).
  Data analyses (multiple logistic regression) will be performed on the cytokine fingerprints of different patient groups taking clinical control of patients into account (sampling during a flare of inflammation versus sampling during disease remission).

SECONDARY OUTCOMES:
Additional measurement of inflammatory cytokines ((interleukin (IL) 1 beta, IL-1RA, IL-6, IL-18, tumor necrosis factor (TNF) alpha, CXCL9 and CXCL10) on serum of patients that are initiated on biological treatment | full study period (up to 48 months)
  In patients included in the study that are initiated on biopharmaceuticals, additional blood sampling will be carried out before start of treatment and after 3 months of therapy. On this blood the FEBRIS Cytokine Profile Assay (measurement of IL-1 beta, IL-1RA, IL-6, IL-18, TNF alpha, CXCL9 and CXCL10) will be performed. The concentration of cytokines will be quantified in pg/ml.
  This data will be used in retrospective analyses with the aim to identify biomarkers or cytokine profiles that separate responders from non-responders.
Registration of age | full study period (up to 48 months)
  At each study visit, the patient's age will be registered through a structured case report form.
  Age will be registered in years or in months if the child is younger than 2 years.
Registration of biological sex | full study period (up to 48 months)
  At each study visit, the patient's biological sex will be registered through a structured case report form.
  Sex will be registered as female, male or intersex
Registration of weight | full study period (up to 48 months)
  At each study visit, the patient's body weight will be registered in kg.
Registration of length | full study period (up to 48 months)
  At each study visit, the patient's length will be registered in cm.
Registration of confirmed or presumed inflammatory diseases | full study period (up to 48 months)
  At each study visit, the patient's known (clinically or genetically confirmed) or tentative inflammatory disease will be registered. This will be registered through a multiple choice list including autoinflammatory disorders (familial Mediterranean fever, tumor necrosis factor receptor associated periodic syndrome, cryopyrin-associated autoinflammatory syndromes, mevalonate kinase deficiency, systemic onset juvenile idiopathic arthritis, periodic fever adenitis pharyngitis and aphthosis, Aicardi-Gutieres syndrome), autoimmune disorders (systemic lupus erythematosus, dermatomyositis, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, oligoarthritic juvenile idiopathic arthritis) or hyperacute inflammatory disease (hemophagocytic lymphohistiocytosis, macrophage activation syndrome, infectious disease related cytokine storm) or other and unspecified inflammatory syndromes.
Registration of clinical symptoms related to inflammatory diseases | full study period (up to 48 months)
  At each study visit, the patient's clinical status will be registered through a multiple-choice list to register the presence or absence of symptoms currently or in the 48 hours before blood sampling. Symptoms include fever, hepatomegaly, splenomegaly, myalgia, arthralgia, exanthema, pharyngitis, oral aphthosis, lymphadenopathy, abdominal pain, thoracic pain, enthesitis.
Registration of current therapy | full study period (up to 48 months)
  At each study visit, the patient's current medication will be registered through a multiple-choice list to register the use of therapeutics that have an effect on inflammation. These include systemic non-steroidal anti-inflammatory drugs, systemic corticosteroids, colchicine, anakinra, canakinumab, tocilizumab, TNF inhibitors, hydroxychloroquine, mycophenolate, methotrexate, janus kinase (JAK) inhibitors, abatacept.
Registration of health-related costs | full study periode (up to 48 months)
  In the subgroup of patients initiated on biopharmaceuticals, health-related costs will be documented.
  To document costs, a questionnaire will be used that was drafted specifically for this project, incorporating registration of the number of visits with caregivers, the type and use of medication, the number and duration of hospitalizations, and questions relating to absence from work.
  A health economic specialist will aggregate the data from this questionnaire to calculate an annual cost in euros per patient.
  This questionnaire will be given to the patients at initiation of biopharmaceutical treatments and every 6 months throughout the study period.
Registration of health-related quality of life | full study periode (up to 48 months)
  In the subgroup of patients initiated on biopharmaceuticals, health-related quality of life (HRQoL) scores will be documented.
  To document HRQoL, the translated version of the PEDsQL and short form 36 (SF-36) will be used for children and adults, respectively.
  The raw scores of PEDsQL are converted into three scale scores: a total score, a psychosocial health score and a physical health score.
  For the SF-36, the item scores are summed into scale scores (weighted sums) and transformed to a 0-100 scale (each question carries equal weight).
  This questionnaire will be given to the patients at initiation of biopharmaceutical treatments and every 6 months throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Filomeen Haerynck, Principal Investigator — University Ghent
Locations (7):
- Belgium (7):
  - UZ Antwerpen, Antwerp
  - ZNA, Antwerp
  - UZ Brussel, Brussels
  - Ghent University Hospital, Ghent
  - UGent, Ghent
  - Jessa Hospital, Hasselt
  - UHasselt, Hasselt

IPD SHARING:
Plan to Share IPD: Yes
raw and anonymized patient clinical and experimental data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: at the end of the study period
Access Criteria: open access